CLINICAL TRIAL: NCT03251131
Title: REstricted Fluid Therapy VERsus Standard trEatment in Acute Kidney Injury - REVERSE-AKI Randomized Controlled Pilot Trial
Brief Title: REVERSE-AKI Randomized Controlled Pilot Trial
Acronym: REVERSE-AKI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Austin Hospital, Melbourne Australia (Other); Guy's and St Thomas' NHS Foundation Trust (Other); University Hospital, Ghent (Other); Medical University Innsbruck (Other); University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Suvi Vaara, MD, PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUS/1782/2017
Record Dates: First submitted 2017-08-12; First posted 2017-08-16 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Acute Kidney Injury; Critical Illness
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restrictive fluid management (Experimental): Restrictive fluid management Targeting a negative or maximum 300ml positive daily fluid balance.
  Interventions: Other: Restrictive fluid management
- Standard therapy (No Intervention): Randomized allocation of standard care at the clinician's discretion in accordance with current best practice.

INTERVENTIONS:
Other: Restrictive fluid management — Daily fluid input is restricted to drugs and nutrition. Fluid boluses and blood products can be given if clinically indicated. Matching fluid output to fluid input whenever possible using diuretics if needed, and additionally, if clinically necessary and plausible, commencing renal replacement therapy. If renal replacement therapy is not deemed clinically desirable, acceptance of a less than targeted fluid balance.
  Arms: Restrictive fluid management

SUMMARY:
Observational studies among patients with acute kidney injury (AKI) have shown an association with fluid accumulation and increased mortality. Trials among other subgroups of critically ill patients have demonstrated that restricting fluid input after the initial resuscitation appears safe.

The objective if this study is to determine whether a fluid restrictive treatment regimen will lead to a lower cumulative fluid balance at 72 hours from randomization in critically ill patients with AKI and whether this approach is safe and feasible.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is common in the critically ill and associates with adverse outcomes. Patients with AKI are frequently have low urine output and are at high risk of developing fluid overload. Fluid overload has been associated with an increased risk for mortality in such patients. Previous trials in critically ill patients found that a 'restrictive fluid therapy' after resuscitation was safe. Implementing a restrictive fluid therapy approach in patients with AKI may also be of benefit. To date, however, no randomized trial has been performed to evaluate the safety and feasibility of implementing a 'restrictive fluid therapy' approach compared to standard fluid therapy in patients with AKI.

In this pilot randomized controlled trial we will evaluate the implementation of a fluid restrictive approach, compared to standard therapy, in adult critically ill patients with acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

1. 18-years or older and admitted to critical care with an arterial line in place
2. The patient has been in critical care for at least 12 hours but no more than 72 hours
3. The patient has AKI but is not receiving acute RRT:

   For the purpose of the study AKI is defined the by the following criteria:
   1. Increase in serum creatinine over 1.5-times above baseline without a decline of 27umol/l or more from the last preceding measurement (at least 12 hours apart) AND/OR
   2. Overall urine output less than 0.5ml/kg/h (or 6ml/kg) for the previous 12h (with urine catheter in place for the period)
4. The patient is judged by the treating clinician not to be intravascularly hypovolemic
5. The patient is likely to remain in critical care for 48 hours after randomization

Exclusion Criteria:

1. Active bleeding necessitating transfusion
2. Maintenance fluid therapy is necessary due to diabetic ketoacidosis, non-ketotic coma, severe burns or other clinical reason determined by the medical staff
3. Need for RRT due to intoxication of a dialyzable toxin
4. Commencement of RRT is expected in the next 6 hours
5. On chronic renal replacement therapy (maintenance dialysis or renal transplant)
6. Presence or a strong clinical suspicion of parenchymal AKI (for example glomerulonephritis, vasculitis, acute interstitial nephritis), or post-renal obstruction
7. Severe hyponatremia (Na <125mmol/L) or hypernatremia (Na >155mmol/L)
8. Need for extracorporeal membrane oxygenation or molecular absorbent recirculating system (MARS-therapy)
9. Pregnant or lactating
10. Patients who are not to receive full active treatment
11. No baseline creatinine available
12. Lack of consent
13. The patient has been enrolled in another trial where co-enrollment is not feasible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Cumulative fluid balance | 72 hours

SECONDARY OUTCOMES:
Duration of acute kidney injury | ICU discharge/14 days
  Defined according to Kidney Disease: Improving Global Outcomes criteria
Number of patients requiring renal replacement therapy | 14 days
Cumulative fluid balance | 24 hours
Cumulative fluid balance | ICU discharge/ 7 days
Cumulative dose of diuretics | ICU discharge/ 7 days

OTHER OUTCOMES:
Number of patients with serious adverse events and reactions | 7 days
  a Ventricular tachycardia/fibrillation b. New onset of atrial fibrillation requiring medication/defibrillation c. Ischemic events i. Acute myocardial infarction ii. Cerebral ischemia verified by CT or MRI scan.
  iii. Intestinal ischemia verified by endoscopy or open surgery.
  iv. Acute peripheral limb ischemia d. Radiologically diagnosed pulmonary edema e. Adverse events related to renal replacement therapy and diuretics use f. Frequency of hypokalaemia (serum K <3.5mmol/L) g. Frequency of hypomagnesaemia (serum Mg <0.8mmol/L) h. frequency of serum pH >7.5 i. other
Mechanical ventilation free days alive | 14 days
Vasopressor free days and alive | 14 days
Renal replacement therapy free days and alive | 90 days
Dialysis dependence | 90 days
All-cause mortality | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Suvi Vaara, MD, PhD, Principal Investigator — Division of Intensive Care Medicine, Department of Anesthesiology, Intensive Care and Pain Medicine, University of Helsinki and Helsinki University Hospital, Helsinki, Finland; Marlies Ostermann, MD, PhD, Principal Investigator — Department of Critical Care and Nephrology, King's College London, Guy's and St Thomas Hospital, Foundation Hospital, London
Locations (7):
- Australia (2):
  - Austin Hospital, Melbourne, Victoria
  - Canberra Hospital, Canberra
- Ghent University Hospital, Ghent, Belgium
- Helsinki University Hospital, Helsinki, Finland
- Lausanne University Hospital, Lausanne, Switzerland
- United Kingdom (2):
  - Guy's and St Thomas Hospital, London
  - Royal London Hospital, Barts Health NHS Trust, London

REFERENCES:
- [Derived] Vaara ST, Ostermann M, Selander T, Bitker L, Schneider A, Poli E, Hoste E, Joannidis M, Zarbock A, van Haren F, Prowle J, Pettila V, Bellomo R. Protocol and statistical analysis plan for the REstricted fluid therapy VERsus Standard trEatment in Acute Kidney Injury-REVERSE-AKI randomized controlled pilot trial. Acta Anaesthesiol Scand. 2020 Jul;64(6):831-838. doi: 10.1111/aas.13557. Epub 2020 Feb 26. PMID 32022904